CLINICAL TRIAL: NCT00492362
Title: A Randomized Controlled Trial of Aerobic Exercise in Patients With End Stage Renal Disease During Outpatient Hemodialysis
Brief Title: Trial of Aerobic Exercise in Patients Undergoing Outpatient Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B2007:067
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Kidney Failure, Chronic
Keywords: hemodialysis; exercise; physical fitness; dialysis adequacy
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Ergometer during hemodialysis
  Interventions: Behavioral: ergometer exercise during hemodialysis
- B (Active Comparator): Pedometer use outside of hemodialysis
  Interventions: Behavioral: pedometer activity outside of hemodialysis

INTERVENTIONS:
Behavioral: ergometer exercise during hemodialysis
  Arms: A
Behavioral: pedometer activity outside of hemodialysis
  Arms: B

SUMMARY:
Randomized controlled trial comparing effects of ergometer exercise during hemodialysis to effects of pedometer use outside of hemodialysis on exercise capacity, functional status, quality of life and adequacy of hemodialysis.

DETAILED DESCRIPTION:
Study Design:

Prospective, randomized, controlled trial of chronic hemodialysis outpatients within the Manitoba Renal Program.

Potential patients include any individual receiving chronic outpatient hemodialysis in Winnipeg (Seven Oaks, Sherbrook, Central and St. Boniface dialysis units) and the Brandon hemodialysis unit.

Exercise Interventions:

Patients will be block randomized to one of the following 2 interventions:

Group A: Cycling on an ergometer GOAL 60 minutes 3 times per week on hemodialysis for 24 weeks A cycling ergometer will be placed on the floor in front of the patient's dialysis chair or at the foot of the bed (if there are only beds available in that unit). The patient will be allowed to exercise anytime during the first half of each dialysis treatment. Goal frequency will be 3 times per week during their usual scheduled hemodialysis treatments.

Group B: Pedometers This group will each receive a pedometer (StepsCount®) at the onset of the study following exercise testing. They will be educated regarding the technical use of the pedometer and will receive the handout entitled "Pedometer Information Sheet: Get Physically Active One Step at a Time!" They will also receive verbal education regarding use of the pedometer and goal activity levels from the exercise study supervisor.

ELIGIBILITY:
Inclusion Criteria:

* All adult (>18 years old) patients
* Treated with hemodialysis for > 3 months
* Hemoglobin > 100 g/L over the previous 2 months
* Kt/V > 1.2 for last month and no history of shortened dialysis due to hemodialysis access issues or frequent alarming during dialysis due to poor access will be eligible for the study.
* Study patients must also be likely able to complete 12 consecutive weeks of exercise (i.e. no travel, change of modality, elective surgery planned) and must be able to comprehend instructions in English.

Exclusion Criteria:

* Acute medical illness in last month
* Unstable hemodialysis with frequent hypotension over the past month
* Active cardiovascular disease (stroke or acute coronary syndrome, unstable angina) in last 3 months
* Lower extremity amputation with no prosthesis (inability to pedal a bike)
* Spine compression fractures
* Severe musculoskeletal pain at rest or with minimal activity
* Inability to sit, stand or walk unassisted (walking devices such as cane will be allowed)
* Shortness of breath at rest or with activities of daily living (NYHA Class IV)
* Labile glycemic control with hypoglycaemic episodes > 1x/week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Aerobic exercise capacity as measured by VO2 peak | 3 and 6 months
physical function as measured by sit to stand to sit; sit and reach and 6 minute walk test | 3 and 6 months

SECONDARY OUTCOMES:
quality of life measured by SF36 | 3 and 6 months
dialysis adequacy as measured by ktV | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clara J Bohm, MD, Principal Investigator — University of Manitoba; Manitoba Renal Program
Locations (4):
- Canada (4):
  - Sherbrook Dialysis Unit, Winnipeg, Manitoba
  - Central Dialysis Unit, Health Sciences Centre, Winnipeg, Manitoba
  - Seven Oaks General Hospital, Winnipeg, Manitoba
  - St. Boniface General Hospital, Winnipeg, Manitoba

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639